CLINICAL TRIAL: NCT05302349
Title: The Effect of Core Stabilization Exercises on Pain Level, Functionality, Stability and Lumbar Multifidus Muscle Cross-sectional Area in People With Chronic Low Back Pain
Brief Title: The Effect of Core Stabilization Exercises in People With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mehmet Akif Guler (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor-Investigator, Mehmet Akif Guler, Lecturer, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-695
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Non-speciﬁc Low Back Pain
Keywords: core exercises; multifidus muscle; lumbar; chronic low back pain; Magnetic resonance imaging; multifidus cross-sectional area

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Outcomes Assessor
Masking Description: The radiologist evaluating the MR images will not know which participant is on which arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Exercise Group (Experimental): Core Exercise Group will performe core stabilization exercises and routine physiotherapy exercises.
  Interventions: Other: Core Exercise Group
- Routine Therapy Group (Active Comparator): Routine Therapy Group will performe routine physiotherapy exercises.
  Interventions: Other: Routine Therapy Group

INTERVENTIONS:
Other: Core Exercise Group — Core Exercise Group Procedure:
  Weeks 1-4 (Five days a week)
  1. Hotpack ultrasound, conventional TENS, stretching exercises and strengthening exercises for low back pain.
  2. Core stabilization exercise :
     * Active pelvic floor exercise (supine position)
     * Bridge exercise (supine position)
     * Back Extension and Ball Back Extension exercises (prone position)
     * Abdominal and Oblique Crunch exercises (supin position)
     * Leg lift exercise (prone position)
     * Plank and Side Plank exercise
     * Superman exercise
  Weeks 5-8 (Three days a week)
  1. Stretching exercises and strengthening exercises for low back pain.
  2. Core stabilization exercise :
     * The same exercises as for Weeks 1-4 will perform.
  Arms: Core Exercise Group
Other: Routine Therapy Group — Routine Therapy Group Procedure:
  Weeks 1-4 (Five days a week)
  1. Hotpack ultrasound, conventional TENS, stretching exercises and strengthening exercises for low back pain.
  Weeks 5-8 (Three days a week)
  1.Stretching exercises and strengthening exercises for low back pain.
  Arms: Routine Therapy Group

SUMMARY:
Low back pain is a health problem that causes clinical, social and economic losses all over the world and affects the majority of the population. More than 80% of adults in the general population experience low back pain at least once in their lifetime. Although the incidence of chronic low back pain is so high, 85% of these pains do not have a pathoanatomical cause and these pains are defined as non-specific chronic low back pain. Exercise therapy is the key to the conservative management of nonspecific chronic low back pain. Lumbar stabilization exercises based on the principle of motor control of core muscles have also become popular in rehabilitation programs for low back pain in recent years.The core region is the lumbopelvic region of the body. The aim of the stabilization exercises is to teach to use the neutral position of the lumbar region and to keep the load on the dynamic and static structures at the lowest level. Core stabilization training begins with teaching the contraction of the transversus abdominus, deep spinal and multifidus muscle.Then, these exercises are planned specifically for the person from immobile positions to movements positions, from simple movements to combined movements, from gross patterns to fine motor patterns, from symmetrical movements to asymmetric movements. These exercises can be developed specifically for the region and pathology with the functions of the muscles in the region of the pathology. The lumbar multifidus muscle is known to be an important stabilizer of the lumbar region. In addition, the cross-sectional area of the lumbar multifidus muscle has short, thick, dense muscle fibers compared to other lumbar region muscles.These dense muscle fibers are compressed in a small space and have a high mass.This morphology allows the lumbar multifidus muscle to produce great force in a small working area and makes the muscle ideal for stability. In addition, the position of the lumbar multifidus muscle between the vertebrae increases its importance for stability. The aim of this study is to determine the effects of core stabilization exercises on the cross-sectional area (CSA) and amount of adipose tissue of the lumbar multifidus muscle in adults with chronic low back pain using magnetic resonance imaging (MRI), and also to examine the effects of these exercises on pain, functionality and lumbopelvic stability.

ELIGIBILITY:
Inclusion Criteria:

* Patient with low back pain for at least 3 months or more
* Age between 18 and 65 years
* Ability to give informed consent

Exclusion Criteria:

* History of previous previous spinal surgery
* Disc herniation with radiculopathy
* Pregnant or breastfeeding
* Systemic disease
* Low back pain due to specific and known causes (Spondylolisthesis, Spinal stenosis, Spondylolysis, Ankylosing spondylitis, Tumor, Structural deformity, Osteoporosis, Rheumatological disease, Infection)
* History of malignancies/cancer
* Unexplained or unintentional weight loss
* Perineal numbness, Bladder dysfunction
* Progressive weakness in lower limbs
* Fracture
* Fever
* Cauda equina syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the amount of adipose tissue and CSA of the muscle by MRI | Baseline - End of the eighth week
  Axial images obtained from the multi-point DIXON (mDIXON) sequence will be used to determine the cross-sectional area and amount of adipose tissue of the lumbar multifidus muscle. The bilateral cross-sectional areas of the lumbar multifidus muscle from the L1-2, L2-3, L3-4, L4-5 and L5-S1 intervertebral disc levels will be calculated by drawing the outlines of the fascial borders of the muscles. Muscle CSA and amount of adipose tissue will be calculated. Subtracting the amount of adipose tissue from the CSA resulting in the functional CSA of the muscle. There will be two measurements, at baseline before the start of program and at the end of the eight weeks intervention.
Visual Analog Scale | Baseline - End of the eighth week
  Pain will be measured using a 10 cm visual analog scale (VAS). Min pain score is 0, max pain score is 10. Participants will mark a point on the VAS that matches the amount of pain they feel.
Oswestry Disability Index | Baseline - End of the eighth week
  Oswestry Disability Index evaluates the extent to which the patient's level of function is restricted by the pain.. Oswestry Disability Index consists of 10 sections, each section the total possible score is ranging from 0 to 5. The score obtained from all questions is added and multiplied by two. The result is noted as a percentage.
  * 0% to 20%= Minimal disability
  * 21% to 40%= Moderate disability
  * 41% to 60%= Severe disability
  * 61% to 80%= Crippling back pain
  * 81% to 100%= Bed-bound or exaggerating symptoms
Sahrmann Core Stability Test | Baseline - End of the eighth week
  The Sahrmann core stability test is a 5-level test used to evaluate the ability of the core muscles to stabilize the spine. While the participant lying in a crook-supine position, the PBU will be inflated to 40 mmHg. Participants will perform the Sahrmann five-level test. A deviation of pressure more than 10 mmHg indicates that the stabilization action of stabilizer muscle has been lost.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Güler, MSc/PT, Principal Investigator — Selcuk University / Faculty of Health Sciences / Department of Physiotherapy and Rehabilitation; Ertuğrul Demirdel, Asst. Prof, Study Chair — Ankara Yildirim Beyazit University / Faculty of Health Sciences / Department of Physiotherapy and Rehabilitation; Ilknur Albayrak Gezer, Assoc. Prof, Study Director — Selcuk University / Faculty of Medicine / Department of Physical Therapy and Rehabilitation; Alaaddin Nayman, Assoc. Prof, Study Director — Selcuk University / Faculty of Medicine / Department of Radiology; Ezgi Akyıldız Tezcan, MD, Study Director — Cumra Public Hospital / Department of Physical Therapy and Rehabilitation
Locations (1):
- Selcuk University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guler MA, Demirdel E, Gezer IA, Nayman A, Tezcan EA. Effect of core stabilization exercises on lumbar multifidus morphology and functional outcomes in chronic non-specific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Dec 28. doi: 10.1186/s12891-025-09433-x. Online ahead of print. PMID 41455992